CLINICAL TRIAL: NCT07048236
Title: Specimen and Clinical Data Collection Plan for LDCT Screening Participants
Status: Recruiting | Type: Observational
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Ministry of Health and Welfare (Ambiguous)
Responsible Party: Principal Investigator, Gee-Chen Chang, Vice president of Chung Shan Medical University, Chung Shan Medical University
Other Study IDs: CS1-25029
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Smoking; Family Relations
Keywords: lung cancer; Low-dose computed tomography; Lung cancer family history; Smoking; proteomic; genomic; Lung cancer risk questionnaire
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, urine samples, lung tissue samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Previous heavy smokers: According to The Lung Cancer Early Detection Program in Taiwan:
  Adults aged 50 to 74 years with a smoking history of at least 20 pack-years, who are either current smokers or have quit smoking within the past 15 years. Current smokers must agree to participate in a smoking cessation program.
  Interventions: Diagnostic Test: Specimen and clinical data collection
- First degree relatives of lung cancer patients: According to The Lung Cancer Early Detection Program in Taiwan:
  Men aged 45 to 74 years and women aged 40 to 74 years who have a biological parent, child, or sibling diagnosed with lung cancer. Individuals who currently smoke must agree to participate in a smoking cessation program.
  Interventions: Diagnostic Test: Specimen and clinical data collection

INTERVENTIONS:
Diagnostic Test: Specimen and clinical data collection — Check total bilirubin, urinary heavy metals,CRP, serum tumor marker, pulmonary function test,Questionnaire

SUMMARY:
Lung cancer remains the leading cause of cancer-related mortality in Taiwan and globally, with increasing incidence and the highest healthcare cost burden among cancers in Taiwan. Despite the widespread use of low-dose computed tomography (LDCT) for screening smokers, over half of lung cancer cases in Taiwan occur in never-smokers, highlighting the need for improved risk stratification. Current national LDCT screening programs do not collect comprehensive risk-related data, limiting their predictive accuracy. This project proposes a five-year, multi-center initiative to establish an integrated biospecimen and clinical data collection system. In its first year, a feasibility pilot will be conducted, followed by recruitment of 12,000 participants. Data collection will include biospecimens (blood, urine, tissue), genomic and proteomic analyses, imaging, and detailed questionnaires covering lifestyle, environmental, and occupational exposures. The project will also develop and validate lung cancer prediction models incorporating epidemiologic, biomarker, air pollution, and imaging data. A Common Data Model (CDM) will be implemented to ensure cross-institutional data standardization and support future international collaboration.

ELIGIBILITY:
Inclusion Criteria:

Previous heavy smokers

According to The Lung Cancer Early Detection Program in Taiwan:

Adults aged 50 to 74 years with a smoking history of at least 20 pack-years, who are either current smokers or have quit smoking within the past 15 years. Current smokers must agree to participate in a smoking cessation program.

First-degree relatives of lung cancer patients

According to The Lung Cancer Early Detection Program in Taiwan:

Men aged 45 to 74 years and women aged 40 to 74 years who have a biological parent, child, or sibling diagnosed with lung cancer. Individuals who currently smoke must agree to participate in a smoking cessation program.

Exclusion Criteria:

1. Pregnancy
2. History of chest computed tomography (including low-dose CT) within the past 12 months.
3. Previous diagnosis of lung cancer
4. Inability to undergo thoracic biopsy or surgery
5. Inability to complete the scan procedure, such as due to being unable to hold their breath.
6. Unexplained hemoptysis within the past month
7. Chest X-ray within the past month showing a clearly suspicious lung lesion
8. Unexplained weight loss exceeding 6 kilograms within the past year

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk population for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-07-17 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Definitive diagnosis of lung lesions confirmed by histopathological or cytological examination. | Measured from time of suspicious imaging finding to histopathological or cytological diagnosis, within a 12 years period

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chung Shan Medical University, Taichung, Taiwan
  - Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City

IPD SHARING:
Plan to Share IPD: No